CLINICAL TRIAL: NCT03954496
Title: Improving Hand Recovery With Neuromodulation in Tetraplegia
Acronym: IGNITE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient study staff
Sponsor: Sara Shahid Salles (Other)
Collaborators: Wings for Life (Other)
Responsible Party: Sponsor-Investigator, Sara Shahid Salles, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201810171642
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injuries; Tetraplegia, Unspecified, Incomplete, Chronic
Keywords: neuroplasticity; rehabilitation; transcranial direct current stimulation; transcranial magnetic stimulation; activities of daily living; motor training
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Bronchiolitis Obliterans Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Experimental): Subjects will receive 20 minutes of active transcranial direct current stimulation at 2.5mA, followed by 2 hours of intensive motor therapy of the more affected upper extremity.
  Interventions: Device: transcranial direct current stimulation; Behavioral: Intensive upper extremity motor training
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of sham transcranial direct current stimulation, followed by 2 hours of intensive motor therapy of the more affected upper extremity.
  Interventions: Device: transcranial direct current stimulation; Behavioral: Intensive upper extremity motor training

INTERVENTIONS:
Device: transcranial direct current stimulation — This is a non-invasive form of stimulation which delivers safe, low levels of electrical current to the brain through the scalp.
Behavioral: Intensive upper extremity motor training — This training is administered one-on-one with an occupational therapist. Activities will be focused on skills the participant wants to regain.

SUMMARY:
This study will examine a form of non-invasive brain stimulation applied with intensive therapy of the arm and hand. The goal of the study is to determine if arm and hand function can be improved in people with incomplete cervical spinal cord injury (neck spinal cord injury, tetraplegia). Participants will be assigned to receive either active or inactive non-invasive brain stimulation.

DETAILED DESCRIPTION:
This study will look at the effects of a painless, non-invasive form of brain stimulation, called transcranial direct current stimulation, or tDCS. tDCS is thought to increase the brain's ability to change. Participants will be assigned to one of two groups by chance. One group will receive tDCS at a level expected to increase the brain's ability to change, while the other group will receive tDCS at a level not thought to affect the brain's ability to change. All participants will receive intensive therapy of their more impaired arm and hand, focusing on exercises that are meaningful to him/her.

ELIGIBILITY:
Inclusion Criteria:

1. traumatic, incomplete cervical SCI sustained at neurological level C4-C7 and classified as B, C or D by the American Spinal Injury Association Impairment Scale (AIS);
2. sustained injury at least 1 year prior to enrollment (i.e., chronic); and
3. Men and women between the ages of 18-65.

Exclusion Criteria:

1. history of head injury, seizures, severe alcohol or drug abuse, or psychiatric illness;
2. cognitive deficits severe enough to preclude informed consent;
3. positive pregnancy test or being of childbearing age and not using appropriate contraception;
4. presence of ferromagnetic material in the cranium except in the mouth, including metal fragments from occupational exposure and surgical clips in or near the brain;
5. decubitus ulcers that might interfere with intervention;
6. cardiac or neural pacemakers;
7. fixed UE contractures;
8. untreated depression;
9. concurrent participation in occupational therapy;
10. within 3 months of recruitment, an addition or change in the dosage of drugs known to exert detrimental effects on motor recovery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Change in Spinal Cord Independence Measure | Change from baseline at immediately post-intervention, 1-month follow-up, 4-month follow-up
  This evaluates self-care, respiration and sphincter management, and mobility.

SECONDARY OUTCOMES:
Change in Medical Research Council Scale Upper Extremity Manual Muscle Test | Change from baseline at immediately post-intervention, 1-month follow-up, 4-month follow-up
  This evaluates the strength of various muscles in the upper extremity. Each muscle that is tested can be scored from a minimum of 0, indicating no strength, up to a maximum of 5, indicating normal strength. Scores are assigned to each side by summing the scores from each of the 41 individual muscles, with a minimum possible total score of 0 and a maximum possible total score of 205. Higher values indicate greater strength.
Change in Canadian Occupational Performance Measure | Change from baseline at immediately post-intervention, 1-month follow-up, 4-month follow-up
  The participant selects 5 tasks they would like to be able to perform, and score their performance as well as satisfaction with their performance of the tasks.
Change in Graded and Redefined Assessment of Strength, Sensibility, and Prehension | Change from baseline at immediately post-intervention, 1-month follow-up, 4-month follow-up
  This measures strength, sensibility, and prehension to obtain information about motor and sensory function.
Change in Van Lieshout Test | Change from baseline at immediately post-intervention, 1-month follow-up, 4-month follow-up
  This test evaluates upper extremity motor performance in cervical spinal cord injury.
Change in cortical motor map volume | Change from baseline at immediately post-intervention, 1-month follow-up, 4-month follow-up
  This is performed using non-invasive transcranial magnetic stimulation to determine which parts of the brain control a muscle in the arm or hand.
Semi-structured interview about study | Baseline
  Participants will be asked about motivations and goals for the study.
Semi-structured interview about study | Immediately post-intervention, 4-month follow-up
  Participants will be asked about their experience in the study, whether they experienced any changes in function during the study, and whether they have recommendations for change.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Salles, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky at Cardinal Hill Rehabilitation Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No